CLINICAL TRIAL: NCT01877213
Title: Coaching of Difficult Diabetic Patients by a Care Coordinating Team After Hospital Discharge
Brief Title: Coaching of Diabetic Patients After Hospital Discharge
Acronym: SORTIDIAB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: P110602; 2012-A00938-35 (Other: IRB number)
Record Dates: First submitted 2013-06-11; First posted 2013-06-13 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2017-04

CONDITIONS: Type 2 Diabetes
Keywords: coaching; therapeutic education; hospital admission; quality improvement strategies; management program; nurse follow up; discharge planning; rehospitalization
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Coaching with coordinate care (Experimental): After discharge from hospital, patients randomized in the coaching group will be coached by a coordinator nurse.
  Interventions: Behavioral: Coaching with coordinate care
- Usual care (No Intervention): After discharge from hospital, patients randomized in the no intervention group will be managed as usually.

INTERVENTIONS:
Behavioral: Coaching with coordinate care — The coordinator nurse will manage ambulatory care with the patient's GP and participate to patient's education.
  Arms: Coaching with coordinate care

SUMMARY:
One third of the costs of medical care for people with diabetes are related to hospitalization." Difficult" diabetic patient, i.e. those with very high HbA1c, patients > 75y, those with diabetic foot ulcers, or those with a recent cardiovascular event have a high rate of readmission when discharged at home after an initial hospitalization related to diabetes or its complications. The objective of the study is to test if a coaching with a care coordinating team after hospital discharge would decrease diabetes-related rehospitalization rate compared with usual care.

DETAILED DESCRIPTION:
Patients with type 1 (T1D) or type 2 diabetes (T2D) hospitalized (>24h) and presenting at least a risk factor for readmission after discharge at home, will be randomized, at time of discharge, between 2 groups: an "intervention" group and a control group (usual management). Intervention will consist in optimized organization of discharge at home followed by a ambulatory individualized coaching by a nurse including an initial situation assessment, a consultation meeting with the patient's GP in order to propose a Health Personalized Plan, then a follow up program with a face to face session each trimester in order to remind the objectives, to assess compliance to the plan, to evaluate difficulties encountered and to help to find solutions. Final data collection will be done in both groups by questioning the patient's general practitioner (GP) and by collecting data on potential hospitalization. Expected duration : 3 years. Readmission rate, duration and causes of hospitalization will be compared between both groups. Impact of the results : Reduction of costs, improved use of hospital specialized resources.

ELIGIBILITY:
Inclusion Criteria:

* type 1 or type 2 diabetes AND AT LEAST ONE of the following criteria:

  * admission for more than 5 days
  * unplanned admission
  * at least one urgent care/emergency room visit in the 6 previous months, whatever its cause
  * HbA1c > 10% on admission
  * cardiovascular event in the previous year : cardiac failure, myocardial infarction, coronary or peripheral revascularization procedure, stage IV peripheral arteriopathy, stroke.
  * occurence during the previous year of a foot lesion requiring an admission or lasting more than one month (foot lesion risk stage 3)

Exclusion Criteria:

* patients with one of the following co-morbidity: cancer in active phase of treatment, Parkinson's disease treated, severe chronic respiratory failure,
* refusal of signing the consent,
* patients non affiliated to Social Security,
* pregnant women,
* people who do not understand French (except if accompanied by somebody able to translate),
* renal dialysis,
* patients aged less than 18 years,
* patients already in a similar type of trial
* the arisen of a pregnancy or a cancer will cause the stop of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2013-06; Primary Completion 2017-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Diabetes-related readmissions | Up to 1 year
  Recording of all readmissions and analysis of files and reports for determining if this readmission was related to diabetes or not.

SECONDARY OUTCOMES:
Causes of rehospitalizations | Up to 1 year
  Each admission to hospital (type of department, duration, direct admission or via Emergency room…) will be recorded. All efforts will be made to record the cause of hospitalization.
Duration of rehospitalizations | Up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Philippe CHANSON, MD, PhD, Principal Investigator — Assistance Publique Hôpitaux de Paris - Bicêtre Hospital
Locations (1):
- Assistance Publique - Hôpitaux de Paris, Bicêtre Hospital, Le Kremlin-Bicêtre, France